CLINICAL TRIAL: NCT03384108
Title: In Vivo Assessment of Glutamine Utilization by Bone Marrow Plasma Cells in Healthy Subjects Using Stable Isotope Resolved Metabolomics: A Pilot Study
Brief Title: In Vivo Assessment of Glutamine Utilization by Bone Marrow Plasma Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wilson I. Gonsalves, M.D., Senior Associate Consultant, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-008291
Record Dates: First submitted 2017-11-03; First posted 2017-12-27 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: In Vivo vs. Ex Vivo assessment of 5-13C-Glutamine incorporation by plasma cells via a bone marrow aspiration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In Vivo (Experimental): Infusion of 5-13C-Glutamine intravenously in healthy subjects prior to undergoing a bone marrow aspiration.
  Interventions: Other: 5-13C-Glutamine; Other: Bone marrow aspiration
- Ex Vivo (Placebo Comparator): Healthy subjects will undergoing a bone marrow aspiration and then the plasma cells acquired will be cultured ex vivo in cell culture media containing 5-13C-Glutamine.
  Interventions: Other: Bone marrow aspiration

INTERVENTIONS:
Other: 5-13C-Glutamine — Intravenous infusion of 5-13C-Glutamine
  Arms: In Vivo
Other: Bone marrow aspiration — Bone marrow aspiration of bone marrow aspirate

SUMMARY:
This pilot study will first establish the feasibility of an in vivo methodology of assessing the utilization of glutamine into the TCA cycle of normal bone marrow plasma cells from healthy subjects while comparing it to an ex vivo approach

DETAILED DESCRIPTION:
Twenty healthy adult study participants between the ages of 18 and 60 years will be recruited to participate in this pilot study that will include two groups: a) Ex Vivo group (10 volunteers) and b) In Vivo group (10 volunteers). Volunteers will be recruited to either group in a sequential alternating fashion.

In vivo 13C SIRM studies evaluating the utilization of glutamine into the TCA cycle of normal bone marrow plasma cells.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* Able to provide written consent

Exclusion Criteria:

* Renal Failure
* Pregnancy
* Active steroid use
* Active liver Disease
* Anemia (Hemoglobin < 12.5 g/dL in men and < 11.5 g/dL in women)
* H/O alcohol use (average > 2 drinks per day)
* BMI > 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of enrichment of 13-Carbon molecules in the TCA cycle metabolites of plasma cells measured by gas chromatography mass spectrometry. | Through study completion, an average of 1 hour
  The plasma cells obtained from the bone marrow aspiration will be processed to determine the percent of 13-carbon enrichment in the various molecules of the TCA cycle within the plasma cells. The outcomes will be reported as a percentage. E.G. 5% of glutamine is labeled with 13-Carbon; e.g. 4% of glutamate is labeled with 13-carbon etc.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Gonsalves, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonsalves WI, Jang JS, Jessen E, Hitosugi T, Evans LA, Jevremovic D, Pettersson XM, Bush AG, Gransee J, Anderson EI, Kumar SK, Nair KS. In vivo assessment of glutamine anaplerosis into the TCA cycle in human pre-malignant and malignant clonal plasma cells. Cancer Metab. 2020 Dec 11;8(1):29. doi: 10.1186/s40170-020-00235-4. PMID 33308307
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials